CLINICAL TRIAL: NCT06905873
Title: A Randomized, Double-Blind, Placebo Controlled, Multi-center Study to Evaluate the Safety and Efficacy of FB102 in Patients With Non-Segmental Vitiligo
Brief Title: A Study to Evaluate the Safety and Efficacy of FB102 in Patients With Non-segmental Vitiligo
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Forte Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FB102-401
Record Dates: First submitted 2025-03-11; First posted 2025-04-02 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Vitiligo
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FB102 (Active Comparator): Participants in this group will receive FB102.
  Interventions: Drug: FB102
- Placebo (Placebo Comparator): Matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: FB102 — Route of administration- Intravenous (IV)
  Arms: FB102
Drug: Placebo — Route of administration- Intravenous (IV)
  Arms: Placebo

SUMMARY:
A Randomized, Double-Blind, Placebo Controlled, Multi-center Study to Evaluate the Safety and Efficacy of FB102 in Patients with Non-Segmental Vitiligo.

DETAILED DESCRIPTION:
Approximately 64 participants who meet all the screening eligibility criteria will be randomized to receive FB102 or placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females aged ≥ 18 to 75 years at time of Screening.
2. Must have confirmed non-segmental vitiligo criteria at the Screening Visit and the Baseline Visit, as assessed by the study investigator.
3. If receiving concomitant medications for any reason other than vitiligo, must be on a stable regimen, which is defined as not starting a new drug or changing dosage within 7 days or 5 half-lives (whichever is longer) prior to Day 1. Participant must be willing to stay on a stable regimen during the duration of the study.

Note: There are additional inclusion criteria. The study center will determine if participant meets all of the criteria

Exclusion Criteria:

1. Currently have active forms of other hypopigmentation (including but not limited to Vogt-Koyanagi-Harada disease, malignancy-induced hypopigmentation [melanoma and mycosis fungoides], post-inflammatory hypopigmentation, pityriasis alba [minor manifestation of atopic dermatitis], senile leukoderma [age-related depigmentation], chemical/drug-induced leukoderma, ataxia telangiectasia, tuberous sclerosis, melasma, and congenital hypopigmentation disorders including piebaldism, Waardenburg syndrome, hypomelanosis of Ito, incontinentia pigmenti, dyschromatosis symmetrica hereditaria, xeroderma pigmentosum, and nevus depigmentosus).
2. Currently have active forms of inflammatory skin disease(s) or evidence of skin conditions (including but not limited to morphea, discoid lupus, leprosy, syphilis, psoriasis, seborrheic dermatitis) at the time of the Screening or Day 1 Visit that in the opinion of the investigator would interfere with evaluation of vitiligo or response to treatment.
3. Greater than approximately 33% leukotrichia (depigmentation of the hair) in areas of vitiligo on the face as assessed by a healthcare professional at the time of screening.

Note: There are additional exclusion criteria. The study center will determine if participant meets all of the criteria

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-emergent adverse events (TEAEs) and Serious Adverse events (SAE) following treatment with FB102 | Upto 16 Weeks post first dose administration
Percent change from Baseline in central read facial-vitiligo area scoring index (F-VASI) | Upto 16 Weeks post first dose administration
  The VASI Score is used to assess the severity and extent of Vitilgo. F-VASI is calculated using a formula that includes involvement of the face (possible range, 0-4), with percentage of vitiligo involvement estimated in finger units by the same investigator throughout the study
Number of participants with percent change from Baseline in central read facial-vitiligo area scoring index (F-VASI) | Upto 16 Weeks post first dose administration
  The VASI Score is used to assess the severity and extent of Vitilgo. F-VASI is calculated using a formula that includes involvement of the face (possible range, 0-4), with percentage of vitiligo involvement estimated in finger units by the same investigator throughout the study

SECONDARY OUTCOMES:
Proportion of participants achieving by percent change improvement in central read F-VASI from Baseline. | Upto 16 Weeks post first dose administration
  The VASI Score is used to assess the severity and extent of Vitilgo. F-VASI is calculated using a formula that includes involvement of the face (possible range, 0-4), with percentage of vitiligo involvement estimated in finger units by the same investigator throughout the study
To evaluate the efficacy of FB102 compared to placebo by percent change from Baseline in total-Vitiligo Area Scoring Index (T-VASI) | Upto 16 Weeks post first dose administration
  T-VASI is calculated using a formula that includes contributions from all body regions (possible range, 0-100). The body is divided into 6 separate and mutually exclusive sites (head/neck, hands, upper extremities [excluding hands], trunk, lower extremities [excluding feet], and feet), with percentage of vitiligo involvement estimated in hand units by the same investigator throughout the study

CONTACTS AND LOCATIONS:
Locations (6):
- Australia (3):
  - Skin & Cancer Foundation Australia - The Skin Hospital, Darlinghurst, New South Wales
  - Novatrials, Kotara, New South Wales
  - Cornerstone Dermatology, Coorparoo, Queensland
- New Zealand (3):
  - Optimal Clinical Trials North, Auckland, Auckland
  - Optimal Clinical Trials Central, Auckland, Auckland
  - Momentum Pukehoke, Auckland, Auckland

IPD SHARING:
Plan to Share IPD: No